CLINICAL TRIAL: NCT03384940
Title: A Phase 2, Multicenter, Open-label Study of DS-8201a in Subjects With HER2-expressing Advanced Colorectal Cancer
Brief Title: DS-8201a in Human Epidermal Growth Factor Receptor2 (HER2)-Expressing Colorectal Cancer (DESTINY-CRC01)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: Daiichi Sankyo (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-J203; 2017-003466-28 (EudraCT Number); 173808 (Registry Identifier: JAPIC CTI); DESTINY-C01 (Other: Daiichi Sankyo and AstraZeneca)
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Neoplasm
Keywords: Oncology; HER2; Colorectal cancer; Antibody drug conjugate; ADC
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DS-8201a Cohort A (Experimental): Cohort A is comprised of participants with HER2-positive (IHC 3+ or IHC 2+/ISH +) who will receive DS-8201a once every 3 weeks
  Interventions: Drug: DS-8201a
- DS-8201a Cohort B (Experimental): Cohort B is comprised of participants with HER2 IHC 2+/ISH - who will receive DS-8201a once every 3 weeks
  Interventions: Drug: DS-8201a
- DS-8201a Cohort C (Experimental): Cohort C is comprised of participants with HER2 IHC 1+ who will receive DS-8201a once every 3 weeks
  Interventions: Drug: DS-8201a

INTERVENTIONS:
Drug: DS-8201a — DS-8201a is comprised of an antibody component conjoined to a drug component in a lyophilized powder, which is made into solution for intravenous administration
  Other Names: Trastuzumab deruxtecan

SUMMARY:
The main objective of this study is to test the safety and effectiveness of DS-8201a for participants with HER2-expressing advanced colorectal cancer.

DETAILED DESCRIPTION:
At study start, only Cohort A is active.

If, and when, Cohort B and C become active depends on the assessment of benefit and risk observed in the program.

The sponsor will inform the investigators if, and when, Cohort B and C are active.

ELIGIBILITY:
Inclusion Criteria:

* Has pathologically documented unresectable, recurrent, or metastatic colorectal adenocarcinoma (until sponsor's notification to the study sites, subject must be a RAS/BRAF wild-type cancer)
* Has received at least 2 prior regimens of standard treatment
* Has measurable disease assessed by the investigator based on RECIST version 1.1.
* Has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1

Exclusion Criteria:

* Has a medical history of myocardial infarction within 6 months, symptomatic congestive heart failure
* Has a medical history of clinically significant lung disease
* Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2020-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (25):
- United States (9):
  - City of Hope Medical Center, Duarte, California
  - University of Southern California, Los Angeles, California
  - UCLA Health, Santa Monica, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Greenville Health System Cancer Institute, Greenville, South Carolina
  - West Cancer Center, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, University of Texas, Houston, Texas
- Italy (4):
  - Università degli studi della Campania L.Vanvitelli, Napoli, Campania
  - Oncology Institute Veneto IOV-IRCCS, Padua, Ferrara
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Lombardo
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan
- Japan (7):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kindai University Hospital, Ōsaka-sayama, Osaka
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-Ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
- Spain (3):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari Clinic de Barcelona, Barcelona
- United Kingdom (2):
  - Royal Marsden Institute (Chelsea), Chelsea, London, England
  - Royal Marsden Institute (Sutton), Sutton, Surrey, England

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Siena S, Raghav K, Masuishi T, Yamaguchi K, Nishina T, Elez E, Rodriguez J, Chau I, Di Bartolomeo M, Kawakami H, Suto F, Koga M, Inaki K, Kuwahara Y, Takehara I, Barrios D, Kobayashi K, Grothey A, Yoshino T. HER2-related biomarkers predict clinical outcomes with trastuzumab deruxtecan treatment in patients with HER2-expressing metastatic colorectal cancer: biomarker analyses of DESTINY-CRC01. Nat Commun. 2024 Nov 25;15(1):10213. doi: 10.1038/s41467-024-53223-3. PMID 39587050
- [Derived] Yoshino T, Di Bartolomeo M, Raghav K, Masuishi T, Loupakis F, Kawakami H, Yamaguchi K, Nishina T, Wainberg Z, Elez E, Rodriguez J, Fakih M, Ciardiello F, Saxena K, Kobayashi K, Bako E, Okuda Y, Meinhardt G, Grothey A, Siena S; DESTINY-CRC01 investigators. Final results of DESTINY-CRC01 investigating trastuzumab deruxtecan in patients with HER2-expressing metastatic colorectal cancer. Nat Commun. 2023 Jun 7;14(1):3332. doi: 10.1038/s41467-023-38032-4. PMID 37286557
- [Derived] Siena S, Di Bartolomeo M, Raghav K, Masuishi T, Loupakis F, Kawakami H, Yamaguchi K, Nishina T, Fakih M, Elez E, Rodriguez J, Ciardiello F, Komatsu Y, Esaki T, Chung K, Wainberg Z, Sartore-Bianchi A, Saxena K, Yamamoto E, Bako E, Okuda Y, Shahidi J, Grothey A, Yoshino T; DESTINY-CRC01 investigators. Trastuzumab deruxtecan (DS-8201) in patients with HER2-expressing metastatic colorectal cancer (DESTINY-CRC01): a multicentre, open-label, phase 2 trial. Lancet Oncol. 2021 Jun;22(6):779-789. doi: 10.1016/S1470-2045(21)00086-3. Epub 2021 May 4. PMID 33961795

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 86 participants who met all inclusion criteria and no exclusion criteria were enrolled and treated at clinic centers in Japan, United States, Spain, and Italy.
Pre-assignment Details: After tissue screening, a total of 86 participants were eligible based on confirmation of HER2 status.
Groups:
- DS-8201a Cohort A: Participants in Cohort A were HER2-positive (IHC 3+ or IHC 2+/ISH +) who received DS-8201a once every 3 weeks.
- DS-8201a Cohort B: Participants in Cohort B were HER2 IHC 2+/ISH - who received DS-8201a once every 3 weeks.
- DS-8201a Cohort C: Participants in Cohort C were HER2/IHC 1+ who received DS-8201a once every 3 weeks.
Period: Overall Study
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Started | 53 | 15 | 18
Completed (As of database lock for final analysis on 28 Dec 2020) | 0 | 0 | 0
Not Completed | 53 | 15 | 18
Not completed — Progressive disease | 36 | 11 | 13
Not completed — Clinical progression | 4 | 0 | 3
Not completed — Adverse Event | 7 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Death | 2 | 1 | 0
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline demographic characteristics were derived from the Full Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C | Total
Number analyzed (Participants) | 53 | 15 | 18 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 8 | 13 | 56
  >=65 years | 18 | 7 | 5 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (11.72) | 61.5 (11.95) | 58.5 (9.97) | 58.4 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 5 | 7 | 40
  Male | 25 | 10 | 11 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 16 | 3 | 8 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 34 | 11 | 8 | 53
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 2 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 10 | 3 | 1 | 14
  Japan | 15 | 3 | 8 | 26
  Italy | 26 | 7 | 8 | 41
  Spain | 2 | 1 | 1 | 4
  United Kingdom | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Best Objective Response Based on Independent Central Review (Confirmed and Unconfirmed) Following DS-8201a Treatment in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Expressing Advanced Colorectal Cancer
Description: Best objective response was reported based on independent central review. As per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1, CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 18 months post-dose
Population: Response was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
Participants
  Confirmed CR | 0 | 0 | 0
  Confirmed PR | 24 | 0 | 0
  Confirmed SD | 20 | 9 | 4
  Confirmed PD | 5 | 5 | 10
  Confirmed Non-evaluable | 4 | 1 | 4
  Unconfirmed CR | 0 | 0 | 0
  Unconfirmed PR | 26 | 0 | 0
  Unconfirmed SD | 18 | 9 | 4
  Unconfirmed PD | 5 | 5 | 10
  Unconfirmed Non-evaluable | 4 | 1 | 4

2. Primary Outcome: Number of Participants With Objective Response Rate Based on Independent Central Review (Confirmed and Unconfirmed) Following DS-8201a Treatment in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Expressing Advanced Colorectal Cancer
Description: Objective response rate (defined as CR+PR) was reported based on independent central review. As per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1, CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: as for outcome 1
Population: Response was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
Participants
  Confirmed CR+PR | 24 | 0 | 0
  Confirmed CR+PR (within 3 months) | 10 | 0 | 0
  Confirmed CR+PR (within 6 months) | 23 | 0 | 0
  Confirmed CR+PR (within 9 months) | 24 | 0 | 0
  Confirmed CR+PR (12 months) | 24 | 0 | 0
  Unconfirmed CR+PR | 26 | 0 | 0
  Unconfirmed CR+PR (within 3 months) | 20 | 0 | 0
  Unconfirmed CR+PR (within 6 months) | 25 | 0 | 0
  Unconfirmed CR+PR (within 9 months) | 25 | 0 | 0
  Unconfirmed CR+PR (within 12 months) | 25 | 0 | 0

3. Secondary Outcome: Number of Participants With Best Objective Response Based on Investigator (Confirmed and Unconfirmed) Following DS-8201a Treatment in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Expressing Advanced Colorectal Cancer
Description: Best objective response was reported based on investigator. As per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1, CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Time Frame: as for outcome 1
Population: Response was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
Participants
  Confirmed CR | 0 | 0 | 0
  Confirmed PR | 25 | 0 | 0
  Confirmed SD | 18 | 7 | 6
  Confirmed PD | 6 | 7 | 8
  Confirmed Non-evaluable | 4 | 1 | 4
  Unconfirmed CR | 0 | 0 | 0
  Unconfirmed PR | 28 | 0 | 0
  Unconfirmed SD | 15 | 7 | 6
  Unconfirmed PD | 6 | 7 | 8
  Unconfirmed Non-evaluable | 4 | 1 | 4

4. Secondary Outcome: Number of Participants With Objective Response Rate Based on Investigator (Confirmed and Unconfirmed) Following DS-8201a Treatment in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Expressing Advanced Colorectal Cancer
Description: Objective response rate (defined as CR+PR) was reported based on investigator. As per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1, CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: as for outcome 1
Population: Response was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
Participants
  Confirmed CR+PR | 25 | 0 | 0
  Unconfirmed CR+PR | 28 | 0 | 0

5. Secondary Outcome: Duration of Response (Confirmed and Unconfirmed) Based on Independent Central Review Following DS-8201a Treatment in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Expressing Advanced Colorectal Cancer
Description: Duration of response (DoR) is defined as the time from the date of the first documentation of an objective response (CR[disappearance of all target lesions] or PR [at least a 30% decrease in the sum of diameters of target lesions]) to the date of the first documentation of PD (at least a 20% increase in the sum of diameters of target lesions). Duration of response was measured for responding participants (CR or PR) only. Month was calculated as (duration of response days × 12)/365.25 for duration of response and calculated as (time to response days × 12)/365.25 for time to response.
Time Frame: Date of first documentation of objective response (CR or PR) up to date of first documentation of PD, up to approximately 18 months post-dose
Population: Duration of response was assessed only in Cohort A in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DS-8201a Cohort A
Number analyzed (Participants) | 53
months
  Confirmed DoR: number analyzed (Participants) | 24
  Confirmed DoR | 7.0 [5.8 to 9.5]
  Unconfirmed DoR: number analyzed (Participants) | 26
  Unconfirmed DoR | 7.0 [5.8 to 9.5]

6. Secondary Outcome: Disease Control Rate (Confirmed and Unconfirmed) Following DS-8201a Treatment in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Expressing Advanced Colorectal Cancer
Description: Disease control rate (DCR) was defined as the proportion of participants who achieved a best overall response of CR + PR + SD based on independent central review and investigator assessment. As per RECIST v1.1, CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions).
Time Frame: as for outcome 1
Population: Duration of response was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
Participants
  Confirmed CR+PR+SD (Independent Central Review) | 44 | 9 | 4
  Unconfirmed CR+PR+SD (Independent Central Review) | 44 | 9 | 4
  Confirmed CR+PR+SD (Investigator) | 43 | 7 | 6
  Unconfirmed CR+PR+SD (Investigator) | 43 | 7 | 6

7. Secondary Outcome: Progression-Free Survival Based on Independent Central Review Following DS-8201a Treatment in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Expressing Advanced Colorectal Cancer
Description: Progression-free survival (PFS) is defined as the time from the date of the first dose to the earlier of the dates of the first objective documentation of radiographic progressive disease (PD) via independent radiologic facility review or death due to any cause. PD was defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Date of first dose to date of first objective documentation of PD or death (whichever occurs first), up to approximately 18 months
Population: Progression-free survival was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
months | 6.9 [4.1 to 8.7] | 2.1 [1.4 to 4.1] | 1.4 [1.3 to 2.1]

8. Secondary Outcome: Progression-Free Survival at Various Time Points Based on Independent Central Review Following DS-8201a Treatment in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Expressing Advanced Colorectal Cancer
Description: Progression-free survival (PFS) is defined as the time from the date of the first dose to the earlier of the dates of the first objective documentation of radiographic progressive disease (PD) via independent radiologic facility review or death due to any cause. PD was defined as at least a 20% increase in the sum of diameters of target lesions.Point estimates at 3, 6, 9, and 12 months are based on Kaplan-Meier estimate. CI is computed using the Brookmeyer-Crowley method. The point estimate percentage (95% confidence interval) at 3, 6, 9, and 12 months is being reported.
Time Frame: as for outcome 7
Population: Progression-free survival was assessed in the Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: point estimate percentage
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
point estimate percentage
  Progression-free survival at 3 months | 74.4 [60.0 to 84.3] | 38.3 [13.0 to 63.6] | 7.5 [0.5 to 28.3]
  Progression-free survival at 6 months | 55 [40.0 to 67.8] | 0 [NA to NA] — Not enough events occurred to estimate the median time or confidence interval. | 0 [NA to NA] — Not enough events occurred to estimate the median time or confidence interval.
  Progression-free survival at 9 months | 34.1 [19.7 to 49.1] | 0 [NA to NA] — Not enough events occurred to estimate the median time or confidence interval. | 0 [NA to NA] — Not enough events occurred to estimate the median time or confidence interval.
  Progression-free survival at 12 months | 19.0 [7.5 to 34.3] | 0 [NA to NA] — Not enough events occurred to estimate the median time or confidence interval. | 0 [NA to NA] — Not enough events occurred to estimate the median time or confidence interval.

9. Secondary Outcome: Overall Survival Based on Independent Central Review Following DS-8201a Treatment in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Expressing Advanced Colorectal Cancer
Description: Overall survival (OS) is defined as the time from the date of first dose to the date of death from any cause.
Time Frame: Time from the date of first dose to date of death from any cause, up to approximately 18 months
Population: Overall survival was assessed in Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
months | 15.5 [8.8 to 20.8] | 7.3 [3.0 to NA] — Not enough events occurred to estimate the confidence interval. | 7.7 [2.2 to 13.9]

10. Secondary Outcome: Overall Survival at Various Time Points Based on Independent Central Review Following DS-8201a Treatment in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Expressing Advanced Colorectal Cancer
Description: Overall survival (OS) is defined as the time from the date of first dose to the date of death from any cause. The point estimate percentage (95% confidence interval) at 3, 6, 9, and 12 months is being reported.
Time Frame: Time from the date of first dose to date of death from any cause, up to approximately 18 months
Population: Overall survival was assessed in Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: point estimate percentage
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
point estimate percentage
  Overall survival at 3 months | 86.8 [74.3 to 93.5] | 86.7 [56.4 to 96.5] | 77.0 [49.7 to 90.7]
  Overall survival at 6 months | 73.6 [59.5 to 83.4] | 53.3 [26.3 to 74.4] | 57.8 [31.0 to 77.3]
  Overall survival at 9 months | 62.0 [47.5 to 73.5] | 38.1 [14.6 to 61.6] | 43.3 [18.9 to 65.7]
  Overall survival at 12 months | 60.0 [45.5 to 71.8] | 38.1 [14.6 to 61.6] | 28.9 [9.3 to 52.3]

11. Secondary Outcome: Pharmacokinetic Parameter Maximum Serum Concentration (Cmax) Following Treatment With DS-8201a in Participants With HER2-expressing Advanced Colorectal Cancer
Description: Maximum serum concentration (Cmax) of DS-8201a and total anti-HER2 antibody was assessed.
Time Frame: Cycle 1: Day 1, before infusion (BI), end of infusion (EOI); Day 8; Day 15; Cycle 2: Day 1, BI and EOI; Cycle 3: Day 1, BI, EOI, 4 hours after start of drug, and 7 hours after start of drug; Cycles 4 and 6: Day 1, BI and EOI
Population: Pharmacokinetic parameters were assessed Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
ug/mL
  DS-8201a | 135 (32.7) | 123 (29.5) | 122 (41.5)
  Total anti-HER2 antibody | 130 (35.1) | 106 (24.6) | 109 (35.4)

12. Secondary Outcome: Pharmacokinetic Parameter Maximum Serum Concentration (Cmax) of MAAA-11181a Following Treatment With DS-8201a in Participants With HER2-expressing Advanced Colorectal Cancer
Description: Maximum serum concentration (Cmax) of MAAA-1181a was assessed.
Time Frame: as for outcome 11
Population: Pharmacokinetic parameters were assessed Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
ng/mL | 15.8 (7.67) | 12.9 (6.40) | 15.1 (5.30)

13. Secondary Outcome: Pharmacokinetic Parameter Time to Maximum Serum Concentration (Tmax) Following Treatment With DS-8201a in Participants With HER2-expressing Advanced Colorectal Cancer
Description: Time to maximum serum concentration (Tmax) of DS-8201a, total anti-HER2 antibody, and MAAA-1181a was assessed.
Time Frame: as for outcome 11
Population: Pharmacokinetic parameters were assessed Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
hours
  DS-8201a | 1.95 [1.42 to 8.75] | 1.72 [1.25 to 5.08] | 3.00 [0.88 to 6.92]
  Total anti-HER2 antibody | 1.72 [1.42 to 6.95] | 1.68 [1.25 to 7.08] | 1.93 [0.88 to 6.92]
  MAAA-1181a | 5.17 [1.75 to 8.75] | 5.00 [3.83 to 6.97] | 5.25 [3.83 to 7.00]

14. Secondary Outcome: Pharmacokinetic Parameter Area Under the Concentration-time Curve (AUC) Following Treatment With DS-8201a in Participants With HER2-expressing Advanced Colorectal Cancer
Description: Area under the concentration-time curve (AUC) from dosing until 21 days (AUC21d) and the last quantifiable concentration (AUClast) of DS-8201a and total anti-HER2 antibody were assessed.
Time Frame: as for outcome 11
Population: Pharmacokinetic parameters were assessed Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug*d/mL
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
ug*d/mL
  DS-8201a: AUC21d: number analyzed (Participants) | 51 | 13 | 16
  DS-8201a: AUC21d | 610 (198) | 571 (208) | 577 (219)
  DS-8201a: AUClast | 600 (204) | 559 (211) | 577 (237)
  Total anti-HER2 antibody: AUC21d: number analyzed (Participants) | 50 | 13 | 16
  Total anti-HER2 antibody: AUC21d | 661 (218) | 569 (224) | 574 (219)
  Total anti-HER2 antibody: AUClast | 638 (235) | 558 (225) | 555 (224)

15. Secondary Outcome: Pharmacokinetic Parameter Area Under the Concentration-time Curve (AUC) of MAAA-1181a Following Treatment With DS-8201a in Participants With HER2-expressing Advanced Colorectal Cancer
Description: Area under the concentration-time curve (AUC) from dosing until 21 days (AUC21d) and the last quantifiable concentration (AUClast) of MAAA-1181a were assessed.
Time Frame: as for outcome 11
Population: Pharmacokinetic parameters were assessed Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*d/mL
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
ng*d/mL
  MAAA-1181a: AUC21d: number analyzed (Participants) | 45 | 12 | 11
  MAAA-1181a: AUC21d | 60.2 (42.7) | 45.0 (28.1) | 55.1 (19.6)
  MAAA-1181a: AUClast | 59.5 (42.1) | 47.1 (29.4) | 62.5 (19.6)

16. Secondary Outcome: Treatment-Emergent Adverse Events (TEAEs) Reported By ≥20% Of Participants Following Treatment With DS-8201a in Participants With HER2-expressing Advanced Colorectal Cancer
Description: A treatment-emergent adverse event (TEAE) is defined as any adverse event not present prior to the initiation of drug treatment or any adverse event already present that worsens in intensity or frequency following exposure to the drug treatment. TEAEs were graded using National Cancer Institute (NCI)-CTCAE version 4.03.
Time Frame: From the date of signing the informed consent form up to 40 (+7) days after last dose, up to approximately 18 months
Population: Adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
Number analyzed (Participants) | 53 | 15 | 18
Participants
  Any TEAE | 53 | 15 | 18
  Nausea | 37 | 9 | 7
  Anaemia | 21 | 4 | 6
  Decreased appetite | 18 | 5 | 7
  Fatigue | 21 | 7 | 3
  Neutrophil count decreased | 20 | 2 | 4
  Platelet count decreased | 17 | 4 | 7
  Vomiting | 23 | 3 | 1
  Diarrhoea | 19 | 0 | 4
  Alopecia | 12 | 4 | 1
  Constipation | 10 | 3 | 1
  Hypokalaemia | 9 | 1 | 4
  Aspartate aminotransferase increased | 6 | 1 | 4
  Malaise | 5 | 0 | 4
  Interstitial lung disease | 4 | 3 | 1
  Dyspnoea | 3 | 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of signing the informed consent form up to 40 (+7) days after last dose, up to approximately 18 months.
Description: A treatment-emergent adverse event (TEAE) was defined as an AE that occurred, having been absent before the first dose of study drug, or having worsened in severity or seriousness after initiation of the study drug until 40 (+7) days after the last dose of the study drug.
Arm/Group | DS-8201a Cohort A | DS-8201a Cohort B | DS-8201a Cohort C
All-Cause Mortality (participants affected / at risk) | 36/53 | 10/15 | 12/18
Serious Adverse Events (participants affected / at risk) | 20/53 | 6/15 | 9/18
Other Adverse Events (participants affected / at risk) | 53/53 | 15/15 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-8201a Cohort A (N=53) | DS-8201a Cohort B (N=15) | DS-8201a Cohort C (N=18)
Sepsis (Infections and infestations) | 3 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Infected fistula (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Meningism (Nervous system disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Disease progression (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Abdominal sepsis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DS-8201a Cohort A (N=53) | DS-8201a Cohort B (N=15) | DS-8201a Cohort C (N=18)
Nausea (Gastrointestinal disorders) | 37 | 9 | 7
Anaemia (Blood and lymphatic system disorders) | 21 | 4 | 6
Decreased appetite (Metabolism and nutrition disorders) | 18 | 5 | 7
Fatigue (General disorders) | 21 | 7 | 3
Neutrophil count decreased (Investigations) | 20 | 2 | 4
Platelet count decreased (Investigations) | 17 | 4 | 7
Vomiting (Gastrointestinal disorders) | 23 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 19 | 0 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 1 | 4
White blood cell count decreased (Investigations) | 11 | 1 | 2
Constipation (Gastrointestinal disorders) | 10 | 3 | 1
Asthenia (General disorders) | 6 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 0
Oedema peripheral (General disorders) | 8 | 1 | 1
Pyrexia (General disorders) | 8 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 6 | 1 | 4
Malaise (General disorders) | 5 | 0 | 4
Alanine aminotransferase increased (Investigations) | 5 | 1 | 3
Blood creatinine increased (Investigations) | 5 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 6 | 2 | 1
Weight decreased (Investigations) | 5 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 2 | 0
Dysgeusia (Nervous system disorders) | 4 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 5 | 0 | 1
Sepsis (Infections and infestations) | 3 | 0 | 1
Urinary tract infection (Infections and infestations) | 5 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 1 | 1
Blood bilirubin increased (Investigations) | 3 | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Hypertension (Vascular disorders) | 3 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Cystitis (Infections and infestations) | 4 | 0 | 0
Gastritis (Gastrointestinal disorders) | 3 | 0 | 0
Haemoglobin decreased (Investigations) | 3 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Disease progression (General disorders) | 1 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 2
Lung infection (Infections and infestations) | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 2 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Blood calcium decreased (Investigations) | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1
Gastrointestinal stoma complication (Gastrointestinal disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal prolapse (Gastrointestinal disorders) | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Dry eye (Eye disorders) | 5 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Blood magnesium decreased (Investigations) | 2 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal sepsis (Gastrointestinal disorders) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Fluid retention (General disorders) | 0 | 0 | 1
Flushing (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Jaundice (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Proctalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Retinal vein occlusion (Vascular disorders) | 0 | 1 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT03384940/Prot_SAP_001.pdf